CLINICAL TRIAL: NCT02318550
Title: A Single Institution Registry Trial Evaluating the Safety of MRI for Patients With Non-MRI Conditional Pacemakers and ICD
Brief Title: Registry of Patients for MRI With Non-MRI Conditional Pacemakers and ICD Non-MRI Conditional Pacemakers and ICD
Status: Completed | Type: Observational
Sponsor: Lancaster General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-68
Record Dates: First submitted 2014-12-10; First posted 2014-12-17 (Estimated); Results first posted 2021-05-17 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: MRI Scans; Magnetic Resonance Imaging; Pacemaker; Implantable Cardioverter Defibrillator
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: MRI Scan — The MRI will be performed with a 1.5 T scanner utilizing institutional protocols and the following settings:
  * Normal operating mode
  * SAR ≤ 2.0 W/kg per patient.

SUMMARY:
The purpose of the registry is to accumulate pre-and post-scan device interrogation data for the purpose of determining the risk of MRI for patients with implantable devices.

DETAILED DESCRIPTION:
Registry Purpose

This registry is a prospective single institution study of MRI examinations in patients with pacemakers or ICD's who will undergo an MRI that is ordered for routine clinical care. The purpose of the registry is to accumulate pre-and post-scan device interrogation data for the purpose of determining the risk of MRI for patients with implantable devices.

Registry data will add to existing data on the safety of MRI scans for patients with pacemakers and ICDs. This safety data may impact physicians' diagnostic choices for this patient population. Patients with conditions for whom MRI is the best diagnostic modality but who have not been able to undergo MRI scanning may be able to do so through registry participation. The diagnostic information obtained from the scan may assist physicians' treatment decisions and may ultimately affect patient outcomes.

In addition, to our knowledge, previous registries of MRI's in non-conditional cardiac devices have been limited to academic centers. This registry would be among the first to demonstrate the feasibility and safety of this approach in a community hospital setting.

Study Methods

The registry research involves acquiring and analyzing the data of device function and adverse events related to the MRI scan.

The need for MRI will be determined on a case-by-case basis based on the patient's medical history and treatment plan/goals, independent of the registry and research purposes. Only patients with implanted devices with orders for clinically indicated MRI scans will be considered for registry inclusion. Clinical review will be performed and the patient considered after determination that no other imaging modality would be appropriate.

The appropriateness of the MRI study must be discussed, in person or via phone call, between a cardiac radiologist, as determined by Paul Leslie, M.D., and the requesting physician. The discussion should include consideration of alternative imaging modalities and diagnostic quality of MRI imaging of requested body region given implanted device(s). The requesting physician is then responsible for discussing with the patient and/or their medical proxy the reasoning for the determination, based on the final decision made by a radiologist.

All patients will be screened prior to enrollment. Any patient with any commercially available pacemaker or ICD system implanted after 2001 who meet all of the inclusion criteria and none of the exclusion criteria, and who require a medically-indicated MRI as described above will be eligible to enroll in the study. The presence/absence of capped/abandoned/epicardial leads/subcutaneous coil will be confirmed and documented by review of the most recent chest x-ray obtained. The x-ray must post-date the most recent device/lead intervention, as determined by a review of the patient's medical record.

If an MRI procedure is deemed absolutely necessary, the MRI will be performed at the Lancaster General Hospital Lime Street MRI facility. MRI scan sequences, field intensity and field(s) of exposure will be selected to minimize risk to the patient while gaining needed diagnostic information for diagnosis or therapy management.

The MRI will be performed with a 1.5 T scanner utilizing institutional protocols and the following settings:

* Normal operating mode
* SAR ≤ 2.0 W/kg per patient.

Prior to the procedure, a pacemaker technologist or manufacturer clinical representative will interrogate the pacemaker or ICD and record the following parameters:

* Patient's underlying rhythm
* Atrial and right/left ventricular pacing thresholds
* P-wave and R-wave amplitude
* Lead impedance (atrial, ventricular, high voltage)
* Battery voltage
* Arrhythmia history
* Tachyarrhythmia therapy

The following pacemaker/ICD parameters will be deactivated for the duration of the MRI:

* Magnet response (ICD)
* Rate response
* PVC response
* Noise reversion response
* Ventricular sense response
* Mode switching
* Tachycardia detection/therapies (ICD)
* EGM triggers

Patients who are not pacemaker dependent will have their pacemaker/ICD programmed to AAI/VVI/DDI at 40 beats per minute for the duration of the MRI. Patients who are pacemaker dependent (pacing at programmed lower rate during the pre-scan interrogation) will have their pacemaker/ICD programmed to AOO/VOO/DOO at the programmed lower rate for the duration of the MRI. Emergency equipment, including a MRI compatible defibrillator and transcutaneous pacemaker, will be available throughout the procedure in the event of an adverse clinical event. In addition to radiology staff, a pacemaker technologist or manufacturer clinical representative and an EP tech/RN with current ACLS will be present for the duration of the procedure. An EP physician/advanced practice provider (APP) must be immediately available (i.e., in the hospital) to provide medical intervention, such as placement of a temporary external pacemaker if required. In the event that a code is called by the MRI staff, hospital protocol indicates that ER staff will respond to the code.

Radiology staff and the electrophysiology (EP) technologist or nurse with current ACLS certification will monitor the following patient parameters at least every 5 minutes throughout the MRI scan:

* Heart rate
* Heart rhythm
* Non-invasive blood pressure
* Oxygen saturation
* Symptoms

If any of the following adverse symptoms/events occur during the scan, the test will be immediately terminated:

* Burning/pulling sensation in device pocket/chest during MRI
* Potentially lethal/previously non-diagnosed arrhythmias during MRI
* Spontaneous and unanticipated pacing rate change
* SOB
* Chest pain
* Feeling of heat/pulling in the chest or device pocket

The patient will be removed from the scanner to the holding area and the device interrogated and reprogrammed to original parameters or as indicated by interrogation. If needed, emergency treatment will be provided as per ACLS protocols or at the discretion of the monitoring physician. The following parameters will be compared to the pre-MRI results:

* Patient's underlying rhythm
* Atrial and right/left ventricular pacing thresholds
* P-wave and R-wave amplitude
* Lead impedance (atrial, ventricular, high voltage)
* Battery voltage

All device-related adverse events/symptoms will be documented on the data collection form and reported to the IRB. The patient will remain in the MRI suite holding area until medically stable. The need for further treatment will be at the discretion of the monitoring physician.

The EP physician/APP will review and compare the pre/post MRI device data prior to the patient's discharge from the MRI suite. Following testing, the pacemaker or ICD will be reprogrammed to the pre-procedure parameters. The need for device reprogramming related to the MRI scan will be based on the clinical judgment of the attending electrophysiologist.

Follow-up

Patients who do not experience any device related adverse events during the MRI will return for one follow-up visit 1-6 weeks after the MRI. The follow-up visit will include pacemaker/ICD interrogation and testing to confirm appropriate function. At a minimum, device interrogation/testing will include:

* Atrial and right/left ventricular pacing thresholds
* P-wave and R-wave amplitude
* Lead impedance (atrial, ventricular, high voltage)
* Battery voltage

Patients who experience one or more device-related adverse events during the MRI will return 1-7 days post-MRI for follow-up pacemaker/ICD testing to confirm appropriate function. At a minimum, device interrogation/testing will include:

* Atrial and right/left ventricular pacing thresholds
* P-wave and R-wave amplitude
* Lead impedance (atrial, ventricular, high voltage)
* Battery voltage

The need for further follow-up will be determined by the physician based on testing results and clinical need.

The results of the follow-up device interrogation, including whether MRI-related adverse events have resolved, will be documented and kept in the device chart and recorded in the Registry database.

If the insurance provider does not cover the MRI and device checks, those costs may be the full responsibility of the patient. The patient will be informed of the status of the pre-authorization before scheduling the MRI.

ELIGIBILITY:
1. Patient has a non-MRI conditional permanently implanted pacemaker or ICD implanted after 2001
2. Patient has a strong clinical indication for MRI where MRI is the diagnostic modality of choice for specific disease state without acceptable alternative imaging technologies as determined by the ordering physician and a radiologist
3. Patient is at least 18 years of age
4. Patient is willing and able to sign study informed consent and HIPAA authorization

Exclusion Criteria:

1. Non-device related contraindication for MRI (such as implanted metallic objects, claustrophobia, morbid obesity)
2. Presence of capped/abandoned/epicardial leads or subcutaneous coil
3. Pregnancy
4. Device generator at elective replacement interval
5. Abdominal device implant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient with any commercially available pacemaker or ICD system implanted after 2001 who meet all of the inclusion criteria and none of the exclusion criteria, and who require a non-cardiac, medically-indicated MRI as described above will be eligible to enroll in the study.
Sampling Method: Non-Probability Sample
Enrollment: 262 (Actual)
Dates: Start 2014-12; Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandeep Bansal, MD, Principal Investigator — Lancaster General Hospital
Locations (1):
- Lancaster General Hospital, Lancaster, Pennsylvania, United States

REFERENCES:
- [Background] Mollerus M, Albin G, Lipinski M, Lucca J. Ectopy in patients with permanent pacemakers and implantable cardioverter-defibrillators undergoing an MRI scan. Pacing Clin Electrophysiol. 2009 Jun;32(6):772-8. doi: 10.1111/j.1540-8159.2009.02364.x. PMID 19545340
- [Background] Nazarian S, Hansford R, Roguin A, Goldsher D, Zviman MM, Lardo AC, Caffo BS, Frick KD, Kraut MA, Kamel IR, Calkins H, Berger RD, Bluemke DA, Halperin HR. A prospective evaluation of a protocol for magnetic resonance imaging of patients with implanted cardiac devices. Ann Intern Med. 2011 Oct 4;155(7):415-24. doi: 10.7326/0003-4819-155-7-201110040-00004. PMID 21969340
- [Background] Nazarian S, Roguin A, Zviman MM, Lardo AC, Dickfeld TL, Calkins H, Weiss RG, Berger RD, Bluemke DA, Halperin HR. Clinical utility and safety of a protocol for noncardiac and cardiac magnetic resonance imaging of patients with permanent pacemakers and implantable-cardioverter defibrillators at 1.5 tesla. Circulation. 2006 Sep 19;114(12):1277-84. doi: 10.1161/CIRCULATIONAHA.105.607655. Epub 2006 Sep 11. PMID 16966586
- [Background] Nazarian S, Beinart R, Halperin HR. Magnetic resonance imaging and implantable devices. Circ Arrhythm Electrophysiol. 2013 Apr;6(2):419-28. doi: 10.1161/CIRCEP.113.000116. No abstract available. PMID 23592868
- [Background] Ferreira AM, Costa F, Tralhao A, Marques H, Cardim N, Adragao P. MRI-conditional pacemakers: current perspectives. Med Devices (Auckl). 2014 May 7;7:115-24. doi: 10.2147/MDER.S44063. eCollection 2014. PMID 24851058
- See also: Magna Safe Registry — http://www.magnasafe.org/aboutmagnasafe.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm: Received MRI: This group received an MRI and pre- and post-imaging device checks.
Period: Overall Study
Arm/Group | Single Arm: Received MRI
Started | 262
Completed | 262
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm: Received MRI
Number analyzed (Participants) | 262
Age, Customized [Mean (Full Range); unit: years]
  Number of participants | 73.9 [39.02 to 101.14]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101
  Male | 161
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 243
  More than one race | 6
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Burning or Pulling Sensations in Chest/Device Pocket During MRI
Time Frame: Through procedure completion, an average of 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm: Received MRI
Number analyzed (Participants) | 262
Participants | 2

2. Primary Outcome: Number of Participants With Potentially Lethal/Previously Non-diagnosed Arrhythmias During MRI
Time Frame: Through procedure completion, an average of 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm: Received MRI
Number analyzed (Participants) | 262
Participants | 0

3. Primary Outcome: Number of Participants With Spontaneous and Unanticipated Pacing Rate Change
Time Frame: Through procedure completion, an average of 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm: Received MRI
Number analyzed (Participants) | 262
Participants | 0

4. Primary Outcome: Number of Participants With Power on Reset of Pacemaker or ICD
Time Frame: Through procedure completion, an average of 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm: Received MRI
Number analyzed (Participants) | 262
Participants | 0

5. Primary Outcome: Number of Participants With MRI Related Device Malfunction/Failure
Time Frame: Through procedure completion, an average of 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm: Received MRI
Number analyzed (Participants) | 262
Participants | 0

6. Primary Outcome: Number of Participants With Serious Injury/Death Related to MRI Device Malfunction/Failure
Time Frame: Through procedure completion, an average of 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm: Received MRI
Number analyzed (Participants) | 262
Participants | 0

7. Primary Outcome: Number of MRI Scans With Post-MRI Device Parameter Change: Greater Than 50 Ohm Change in Atrial or Ventricular (RV and/or LV) Lead Impedance
Time Frame: Through procedure completion, an average of 1 hour
Measure: Count of Units; unit: MRI Scan
Units Other Than Participants: MRI Scan
Arm/Group | Single Arm: Received MRI
Number analyzed (Participants) | 262
Number analyzed (MRI Scan) | 318
MRI Scan | 19

8. Primary Outcome: Number of MRI Scans With Post-MRI Device Parameter Changes: Greater Than 5 Ohm Change in High Voltage Lead Impedance
Time Frame: Through procedure completion, an average of 1 hour
Measure: Count of Units; unit: MRI Scan
Units Other Than Participants: MRI Scan
Arm/Group | Single Arm: Received MRI
Number analyzed (Participants) | 262
Number analyzed (MRI Scan) | 318
MRI Scan | 1

9. Primary Outcome: Number of MRI Scans With Post-MRI Device Parameter Changes: Greater Than 50% Decrease in Atrial or Ventricular (RV and/or LV) Sensing Threshold
Time Frame: Through procedure completion, an average of 1 hour
Measure: Count of Units; unit: MRI Scan
Units Other Than Participants: MRI Scan
Arm/Group | Single Arm: Received MRI
Number analyzed (Participants) | 262
Number analyzed (MRI Scan) | 318
MRI Scan | 0

10. Primary Outcome: Number of MRI Scans With Post-MRI Device Parameter Changes: Greater Than or Equal to a 1 Volt Increase in Atrial or Ventricular (RV and/or LV) Pacing Threshold
Time Frame: Through procedure completion, an average of 1 hour
Measure: Count of Units; unit: MRI Scan
Units Other Than Participants: MRI Scan
Arm/Group | Single Arm: Received MRI
Number analyzed (Participants) | 262
Number analyzed (MRI Scan) | 318
MRI Scan | 0

ADVERSE EVENTS:
Time Frame: up to 1 hour following MRI
Arm/Group | Single Arm: Received MRI
All-Cause Mortality (participants affected / at risk) | 0/262
Serious Adverse Events (participants affected / at risk) | 0/262
Other Adverse Events (participants affected / at risk) | 4/262
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm: Received MRI (N=262)
Burning/pulling sensation (Product Issues) | 3 (3) — Burning/pulling sensation in device pocket/chest during MRI
Chest Pain (Cardiac disorders) | 1 (1) — Pain in chest during MRI

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-17): https://cdn.clinicaltrials.gov/large-docs/50/NCT02318550/Prot_SAP_000.pdf